CLINICAL TRIAL: NCT05111548
Title: Neuromodulation Plus Cognitive Training to Improve Working Memory Among Individuals With Severe Mental Illness
Brief Title: Brain Stimulation and Cognitive Training - Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cynthia Burton, Clinical Assistant Professor, Department of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00119204b
Record Dates: First submitted 2021-10-01; First posted 2021-11-08 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active stimulation + cognitive training (Experimental): Participants receive 10 sessions of 'active' non-invasive brain stimulation (tDCS) with concurrent cognitive training (BrainHQ).
  Interventions: Device: tDCS (Active); Behavioral: BrainHQ
- Inactive stimulation + cognitive training (Sham Comparator): Participants receive 10 sessions of 'inactive' non-invasive brain stimulation (tDCS) with concurrent cognitive training (BrainHQ).
  Interventions: Behavioral: BrainHQ; Device: tDCS (Inactive)

INTERVENTIONS:
Device: tDCS (Active) — tDCS is a non-invasive procedure in which electrodes are attached to the scalp and send a small direct current to stimulate brain function. Participants in the experimental arm will receive a steady current delivery through the device.
  Other Names: transcranial direct current stimulation
  Arms: Active stimulation + cognitive training
Behavioral: BrainHQ — BrainHQ is a web-based, commercially available cognitive training program that includes exercises to enhance working memory
  Other Names: cognitive training; computerized cognitive exercises
Device: tDCS (Inactive) — tDCS is a non-invasive procedure in which electrodes are attached to the scalp and send a small direct current to stimulate brain function. Participants in the sham arm will wear the device but will not receive a steady current delivery.
  Other Names: transcranial direct current stimulation
  Arms: Inactive stimulation + cognitive training

SUMMARY:
People with serious mental illness often experience difficulties with thinking skills like memory. These difficulties can make it harder to perform day-to-day activities. The purpose of this study is to test whether combining a type of non-invasive brain stimulation with computerized cognitive exercises is helpful in improving a specific type of memory skill in people who have mental health conditions.

The study is a randomized clinical trial, meaning that participants will be randomly assigned to receive either 'active' or 'inactive' brain stimulation. All participants will complete computerized cognitive exercises, also known as cognitive training.

Overall, participants will be in the study for 6-8 weeks. The study involves 10 visits to the clinic over 2-4 weeks for cognitive training and either active or inactive brain stimulation. Participants will also complete paper-and-pencil assessments at the beginning and end of treatment, and one month after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder I or II, schizoaffective disorder, or schizophrenia
* Willingness to participate in study procedures

Exclusion Criteria:

* History of neurological illness or injury (e.g., stroke)
* History of loss of consciousness
* Diagnosed intellectual disability
* Current substance use disorder
* Current mania or moderate depression or severe psychosis
* Current serious suicidal ideation/behavior
* Pregnant or trying to become pregnant, or currently lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Burton, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants did not meet the inclusion criteria and were excluded from further participation (i.e., screen failures). Two participants withdrew from the study after enrollment and prior to randomization. Therefore, 19 participants were enrolled and 15 were assigned.
Period: Overall Study
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
Started | 8 | 7
Completed | 5 | 6
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.63 (8.43) | 34.71 (11.43) | 33.07 (9.70)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender Identity
  Participants
    Woman | 4 | 5 | 9
    Man | 3 | 2 | 5
    Non-binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15
MCCB spatial span total score [Mean (Standard Deviation); unit: points on a scale] — Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) spatial span total raw score. Spatial span is a subtest of the standardized MCCB and a measure of visual working memory. Examinees must tap sequences of blocks in the same order as the examiner then in reverse. Correct responses are summed for the forward and backward condition to create a total raw score (0-32, where higher scores indicate better performance).
  points on a scale | 17.25 (2.87) | 15.57 (4.65) | 16.47 (3.76)
MCCB letter-number span total score [Mean (Standard Deviation); unit: points on a scale] — Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) letter-number span total raw score. Letter-number span is a subtest of the standardized MCCB and a measure of verbal working memory. Examinees must reorder sequences of numbers and letters spoken out loud by the examiner. Correct responses are counted to create a total score (0-24, where higher scores indicate better performance).
  points on a scale | 15.38 (3.38) | 15.43 (3.60) | 15.40 (3.36)
MCCB Trail Making Test, part A [Mean (Standard Deviation); unit: seconds] — MCCB Trail Making Test, part A. The Trail Making Test, part A is a subtest of the standardized MCCB and a measure of visuomotor processing/sequencing speed. Examinees must draw a line connecting numbers in ascending order as quickly as possible. Completion time in seconds is recorded (0-120, where lower scores represent better performance).
  seconds | 22.50 (6.09) | 23.14 (4.98) | 22.80 (5.41)
Trail Making Test, part B [Mean (Standard Deviation); unit: seconds] — Trail Making Test, part B is not part of the standardized MCCB, but is commonly administered alongside part A as a measure of speeded visuomotor switching/flexibility. Examinees must draw a line connecting numbers and letters in alternating order (e.g., 1-A-2-B). Completion time in seconds is recorded (0-300, where lower scores represent better performance).
  seconds | 60.50 (11.67) | 72.71 (24.94) | 66.20 (19.35)

OUTCOME MEASURES:

1. Primary Outcome: Change in Working Memory Performance - Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Letter-number Span Total Score
Description: MCCB letter-number span total raw score. Letter-number span is a subtest of the standardized MCCB and a measure of verbal working memory. Examinees must reorder sequences of numbers and letters spoken out loud by the examiner. Correct responses are counted to create a total score (0-24, where higher scores indicate better performance). For change scores, a positive value indicates improvement (i.e., higher total score).
Time Frame: Baseline to post-treatment (up to 4 weeks)
Population: Four participants withdrew from the study before post-treatment assessment and were not included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
Number analyzed (Participants) | 5 | 6
score on a scale | 0.40 (1.67) | 0.50 (1.64)
Statistical Analysis 1: Comparison: Active Stimulation + Cognitive Training vs Inactive Stimulation + Cognitive Training; Mixed ANOVA (within-subjects factor=time; between-subjects factor=group); Test type: Superiority; p = 0.923, ANOVA

2. Primary Outcome: Change in Working Memory Performance - Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Spatial Span Total Score
Description: MCCB spatial span total raw score. Spatial span is a subtest of the standardized MCCB and a measure of visual working memory. Examinees must tap sequences of blocks in the same order as the examiner then in reverse. Correct responses are summed for the forward and backward condition to create a total raw score (0-32, where higher scores indicate better performance).For change scores, a positive value indicates improvement (i.e., higher total score).
Time Frame: Baseline to post-treatment (up to 4 weeks)
Population: Four participants withdrew from the study before post-treatment assessment and were not included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
Number analyzed (Participants) | 5 | 6
score on a scale | 1.60 (0.89) | 0.17 (1.60)
Statistical Analysis 1: Comparison: Active Stimulation + Cognitive Training vs Inactive Stimulation + Cognitive Training; Mixed ANOVA (within-subjects factor=time; between-subjects factor=group); Test type: Superiority; p = 0.110, ANOVA

3. Secondary Outcome: Change in Non-Working Memory Comparison Measures - MCCB Trail Making Test, Part A
Description: The Trail Making Test, part A is a subtest of the standardized MCCB and a measure of visuomotor processing/sequencing speed. Examinees must draw a line connecting numbers in ascending order as quickly as possible. Completion time in seconds is recorded (0-120, where lower scores represent better performance). For change scores, a positive value indicates improvement (i.e., faster completion time).
Time Frame: Baseline to post-treatment (up to 4 weeks)
Population: Four participants withdrew from the study before post-treatment assessment and were not included in the analyses.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
Number analyzed (Participants) | 5 | 6
seconds | 1.40 (5.55) | 2.33 (7.17)
Statistical Analysis 1: Comparison: Active Stimulation + Cognitive Training vs Inactive Stimulation + Cognitive Training; Mixed ANOVA (within-subjects factor=time; between-subjects factor=group); Test type: Superiority; p = 0.818, ANOVA

4. Secondary Outcome: Change in Non-Working Memory Comparison Measures - Trail Making Test, Part B
Description: Trail Making Test, part B is not part of the standardized MCCB, but is commonly administered alongside part A as a measure of speeded visuomotor switching/flexibility. Examinees must draw a line connecting numbers and letters in alternating order (e.g., 1-A-2-B). Completion time in seconds is recorded (0-300, where lower scores represent better performance). For change scores, a positive value indicates improvement (i.e., faster completion time).
Time Frame: Baseline to post-treatment (up to 4 weeks)
Population: Four participants withdrew from the study before post-treatment assessment and were not included in the analyses.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
Number analyzed (Participants) | 5 | 6
seconds | 3.60 (12.82) | 19.50 (17.76)
Statistical Analysis 1: Comparison: Active Stimulation + Cognitive Training vs Inactive Stimulation + Cognitive Training; Mixed ANOVA (within-subjects factor=time; between-subjects factor=group); Test type: Superiority; p = 0.130, ANOVA

ADVERSE EVENTS:
Time Frame: Duration of participation in the study (i.e., up to 8 weeks).
Arm/Group | Active Stimulation + Cognitive Training | Inactive Stimulation + Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation + Cognitive Training (N=8) | Inactive Stimulation + Cognitive Training (N=7)
Intense discomfort at stimulation site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05111548/Prot_SAP_000.pdf